CLINICAL TRIAL: NCT06046794
Title: Phase IV Study Assessing Efficacy of First-Line Chemotherapy With Gemcitabine in GemCore+ Metastatic Pancreatic Adenocarcinoma Patients Ineligible to FOLFIRINOX Treatment
Brief Title: Efficacy of First-Line Gemcitabine Chemotherapy in GemCore+ Metastatic Pancreatic Adenocarcinoma Patients
Acronym: GemSign-01
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GemSign-01-IPC 2022-068
Record Dates: First submitted 2023-09-06; First posted 2023-09-21 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Cancer Of Pancreas
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- metastatic pancreatic adenocarcinoma patients (Experimental): Analyze of GemCore status
  Interventions: Other: Analyze of GemCore status

INTERVENTIONS:
Other: Analyze of GemCore status — Genomic analyze of GemCore status

SUMMARY:
The goal of this interventional study is to learn about the efficacy of first-line chemotherapy with Gemcitabine in metastatic pancreatic adenocarcinoma patients expressing the GemCore signature in their tumor. The main question it aims to answer is to assess efficacy of Gemcitabine (tumor response, survival rate) in the population of patient bearing the GemCore signature.

Participants will start the chemotherapy with Gemcitabine as usually performed in standard care of their center. They will consent to a genomic analyze of their tumor to know if it bears the GemCore signature. The center will manage the participant's follow up as usually realized in standard care.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic pancreatic adenocarcinoma histological proved
* FOLFIRINOX chemotherapy-ineligible patient and going to receive first-line metastatic chemotherapy with gemcitabine monotherapy
* Tumor material allowing assessment of GEMCore status (i.e. FFPE block with tumor cellularity ≥ 10%);
* Life expectancy > 2 months;
* Measurable target according to RECIST 1.1 criteria;
* No previous treatment in metastatic situation;
* Age ≥ 18 years;
* Patient not opposed to study participation;
* Affiliation to a social security system, or beneficiary of such a scheme.

Exclusion Criteria:

* Contraindication to Gemcitabine treatment;
* ECOG performance status ≥ 3;
* Person in emergency situation or unable to express non-opposition;
* Patient under a legal protection measure (adult under guardianship, curatorship or safeguard of justice);
* Unable to undergo medical follow-up for geographical, social or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of alive GemCore+ patients treated with Gemcitabine | 12 months
  Percentage of alive GemCore+ patients treated with Gemcitabine

SECONDARY OUTCOMES:
Overall survival | 24 months
  Overall survival
Tumor response rate | 24 months
  Tumor response rate
Progression-free survival | 24 months
  Progression-free survival

OTHER OUTCOMES:
Overall survival of GemCore- patients | 24 months
  Overall survival of GemCore- patients

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Paoli Calmettes, Marseille, France

IPD SHARING:
Plan to Share IPD: No